CLINICAL TRIAL: NCT00930761
Title: A Randomized Controlled Trial to Evaluate the Effects of Music Therapy on Breastfeeding Rates Among Mothers of Premature Newborns
Brief Title: Effects of Music Therapy on Breastfeeding Among Mothers of Premature Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Maternidade Escola da UFRJ (Unknown); Instituto de Puericultura e Pediatria Martagão Gesteira (Unknown)
Responsible Party: Arnaldo P Barbosa, Department of Pediatris, UFRJ School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAME-21-2001
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Breastfeeding
Keywords: breast feeding; music therapy; maternal welfare; infant, newborn
MeSH Terms: conditions — Breast Feeding | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Music therapy (Experimental)
  Interventions: Behavioral: Music therapy

INTERVENTIONS:
Behavioral: Music therapy — Music therapy sessions systematically offered to all mothers in the intervention group, three times a week, not mandatory, conducted by two music therapists in an appropriate room, during 60 minutes.
  Other Names: MT
  Arms: Music therapy

SUMMARY:
The purpose of this study is to evaluate the impact of music therapy on breastfeeding rates among mothers of premature newborns.

Hypothesis: Music therapy applied to mothers of premature newborns increases the rates of maternal breastfeeding at the time of the infant hospital discharge and at follow-up visits.

DETAILED DESCRIPTION:
Music therapy has been shown to have positive effects in several areas such as mental health, special education, rehabilitation and social development. Its use as a means to facilitate communication and expression of emotional contents was shown to be able to promote relief of anxiety, fears and tensions. However, in the maternal and child health area there are still few studies demonstrating the contribution of this therapy in the promotion of health and no study evaluating specifically the impact of this intervention on the rates of breastfeeding in mothers of premature newborns.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of premature newborns, with birth weight ≤ 1750 g that have reached clinical stability defined by the medical staff.
* To have signed an informed consent to participate in the study.

Exclusion Criteria:

* Mothers that are HIV (Human Immunodeficiency Virus) positive.
* Mothers of neonates with clinical problems that impaired breast suction (encephalopathy with serious hypotonus, oro-facial anomalies, and heart problems).
* Mothers with severe hearing deficiencies.

Exit Criteria:

* Mothers whose neonates died during the hospital stay.
* Mothers who, for any reason, had three or less music therapy sessions.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2004-03; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha NS Vianna, MSc, Principal Investigator — UFRJ (Universidade Federal do Rio de Janeiro) Maternidade Escola; Arnaldo P Barbosa, MD, MSc, PhD, Study Director — UFRJ School of Medicine, Department of Pediatrics; Albelino S Carvalhaes, Study Chair — UFRJ Maternidade Escola; Antonio LA Cunha, MD, MSc, PhD, Study Chair — UFRJ School of Medicine, Department of Pediatrics
Locations (1):
- UFRJ Maternidade Escola, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Al-Qahtani NH. Foetal response to music and voice. Aust N Z J Obstet Gynaecol. 2005 Oct;45(5):414-7. doi: 10.1111/j.1479-828X.2005.00458.x. PMID 16171479
- [Background] Arnon S, Shapsa A, Forman L, Regev R, Bauer S, Litmanovitz I, Dolfin T. Live music is beneficial to preterm infants in the neonatal intensive care unit environment. Birth. 2006 Jun;33(2):131-6. doi: 10.1111/j.0730-7659.2006.00090.x. PMID 16732778
- [Background] Barrera ME, Rykov MH, Doyle SL. The effects of interactive music therapy on hospitalized children with cancer: a pilot study. Psychooncology. 2002 Sep-Oct;11(5):379-88. doi: 10.1002/pon.589. PMID 12228871
- [Background] Berbel P, Moix J, Quintana S. [Music versus diazepam to reduce preoperative anxiety: a randomized controlled clinical trial]. Rev Esp Anestesiol Reanim. 2007 Jun-Jul;54(6):355-8. Spanish. PMID 17695946
- [Background] Caine J. The effects of music on the selected stress behaviors, weight, caloric and formula intake, and length of hospital stay of premature and low birth weight neonates in a newborn intensive care unit. J Music Ther. 1991 Winter;28(4):180-92. doi: 10.1093/jmt/28.4.180. PMID 10160836
- [Background] Caprilli S, Anastasi F, Grotto RP, Scollo Abeti M, Messeri A. Interactive music as a treatment for pain and stress in children during venipuncture: a randomized prospective study. J Dev Behav Pediatr. 2007 Oct;28(5):399-403. doi: 10.1097/DBP.0b013e31811ff8a7. PMID 18049324
- [Background] Chang MY, Chen CH, Huang KF. Effects of music therapy on psychological health of women during pregnancy. J Clin Nurs. 2008 Oct;17(19):2580-7. doi: 10.1111/j.1365-2702.2007.02064.x. Epub 2008 Feb 19. PMID 18298503
- [Background] Chou LL, Wang RH, Chen SJ, Pai L. Effects of music therapy on oxygen saturation in premature infants receiving endotracheal suctioning. J Nurs Res. 2003 Sep;11(3):209-16. doi: 10.1097/01.jnr.0000347637.02971.ec. PMID 14579198
- [Background] Clark ME, McCorkle RR, Williams SB. Music therapy-assisted labor and delivery. J Music Ther. 1981 Summer;18(2):88-100. doi: 10.1093/jmt/18.2.88. PMID 10252815
- [Background] Desquiotz-Sunnen N. [Singing for preterm born infants music therapy in neonatology]. Bull Soc Sci Med Grand Duche Luxemb. 2008;Spec No 1:131-43. French. PMID 18404877
- [Background] Ferrer AJ. The effect of live music on decreasing anxiety in patients undergoing chemotherapy treatment. J Music Ther. 2007 Fall;44(3):242-55. doi: 10.1093/jmt/44.3.242. PMID 17645387
- [Background] Jones G, Steketee RW, Black RE, Bhutta ZA, Morris SS; Bellagio Child Survival Study Group. How many child deaths can we prevent this year? Lancet. 2003 Jul 5;362(9377):65-71. doi: 10.1016/S0140-6736(03)13811-1. PMID 12853204
- [Background] Hatem TP, Lira PI, Mattos SS. The therapeutic effects of music in children following cardiac surgery. J Pediatr (Rio J). 2006 May-Jun;82(3):186-92. doi: 10.2223/JPED.1473. Epub 2006 May 4. PMID 16680285
- [Background] Klassen JA, Liang Y, Tjosvold L, Klassen TP, Hartling L. Music for pain and anxiety in children undergoing medical procedures: a systematic review of randomized controlled trials. Ambul Pediatr. 2008 Mar-Apr;8(2):117-28. doi: 10.1016/j.ambp.2007.12.005. PMID 18355741
- [Background] Krout RE. The effects of single-session music therapy interventions on the observed and self-reported levels of pain control, physical comfort, and relaxation of hospice patients. Am J Hosp Palliat Care. 2001 Nov-Dec;18(6):383-90. doi: 10.1177/104990910101800607. PMID 11712719
- [Background] Lai HL, Chen CJ, Peng TC, Chang FM, Hsieh ML, Huang HY, Chang SC. Randomized controlled trial of music during kangaroo care on maternal state anxiety and preterm infants' responses. Int J Nurs Stud. 2006 Feb;43(2):139-46. doi: 10.1016/j.ijnurstu.2005.04.008. Epub 2005 Jul 5. PMID 15996669
- [Background] Liu RW, Mehta P, Fortuna S, Armstrong DG, Cooperman DR, Thompson GH, Gilmore A. A randomized prospective study of music therapy for reducing anxiety during cast room procedures. J Pediatr Orthop. 2007 Oct-Nov;27(7):831-3. doi: 10.1097/BPO.0b013e3181558a4e. PMID 17878794
- [Background] Phumdoung S, Good M. Music reduces sensation and distress of labor pain. Pain Manag Nurs. 2003 Jun;4(2):54-61. doi: 10.1016/s1524-9042(02)54202-8. PMID 12836149
- [Background] Standley JM, Moore RS. Therapeutic effects of music and mother's voice on premature infants. Pediatr Nurs. 1995 Nov-Dec;21(6):509-12, 574. PMID 8700604
- [Background] Victora CG, Wagstaff A, Schellenberg JA, Gwatkin D, Claeson M, Habicht JP. Applying an equity lens to child health and mortality: more of the same is not enough. Lancet. 2003 Jul 19;362(9379):233-41. doi: 10.1016/S0140-6736(03)13917-7. PMID 12885488
- [Background] Wong HL, Lopez-Nahas V, Molassiotis A. Effects of music therapy on anxiety in ventilator-dependent patients. Heart Lung. 2001 Sep-Oct;30(5):376-87. doi: 10.1067/mhl.2001.118302. PMID 11604980
- [Background] Emery CF, Hsiao ET, Hill SM, Frid DJ. Short-term effects of exercise and music on cognitive performance among participants in a cardiac rehabilitation program. Heart Lung. 2003 Nov-Dec;32(6):368-73. doi: 10.1016/s0147-9563(03)00120-1. PMID 14652528
- [Background] Hilliard RE. The effects of music therapy on the quality and length of life of people diagnosed with terminal cancer. J Music Ther. 2003 Summer;40(2):113-37. doi: 10.1093/jmt/40.2.113. PMID 14505443
- [Background] Nilsson U, Rawal N, Unosson M. A comparison of intra-operative or postoperative exposure to music--a controlled trial of the effects on postoperative pain. Anaesthesia. 2003 Jul;58(7):699-703. doi: 10.1046/j.1365-2044.2003.03189_4.x. PMID 12886915
- [Background] Yilmaz E, Ozcan S, Basar M, Basar H, Batislam E, Ferhat M. Music decreases anxiety and provides sedation in extracorporeal shock wave lithotripsy. Urology. 2003 Feb;61(2):282-6. doi: 10.1016/s0090-4295(02)02375-0. PMID 12597931
- [Background] Hamel WJ. The effects of music intervention on anxiety in the patient waiting for cardiac catheterization. Intensive Crit Care Nurs. 2001 Oct;17(5):279-85. doi: 10.1054/iccn.2001.1594. PMID 11866419
- [Background] Lepage C, Drolet P, Girard M, Grenier Y, DeGagne R. Music decreases sedative requirements during spinal anesthesia. Anesth Analg. 2001 Oct;93(4):912-6. doi: 10.1097/00000539-200110000-00022. PMID 11574356
- See also: American Music Therapy Association — http://www.musictherapy.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 03/01/2004 to 07/31/2007. Mothers of LBW newborns (≤ 1750g) that have reached clinical stability and signed an informed consent.
Pre-assignment Details: Eligible mothers: 190. Excluded: 89 (26 because their neonates fullfiled one of the exclusion criteria, 18 because their newborns died before being considered in clinical stability, 11 because they did not agree to participate and 34 because they could not be accessed during the newborn hospital stay, most for receiving early hospital discharge).
Period: Overall Study
Arm/Group | Control | Music Therapy
Started | 50 | 51
Completed | 46 | 48
Not Completed | 4 | 3
Not completed — 3 newborns died; 1 mother quit the study | 4 | 0
Not completed — less than 3 music therapy sessions | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Music Therapy | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Customized [Number; unit: participants] — 12-20 years; 21-30 years; 31-40 years; > 40 years
  participants
    12-20 years | 13 | 13 | 26
    21-30 years | 22 | 27 | 49
    31-40 years | 12 | 9 | 21
    > 40 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 101
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Maternal Breastfeeding at Infant Discharge
Description: Maternal breastfeeding means exclusive maternal breastfeeding, predominant maternal breastfeeding (maternal milk associated to other liquid, except formula) and continuous maternal breastfeeding (maternal milk associate to other food, including formula).
Time Frame: At the time of the infant hospital discharge
Population: Analysis by intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 46 | 48
participants | 33 | 42
Statistical Analysis 1: Comparison: Control vs Music Therapy; Null hypothesis: Music therapy does not increase the rate of maternal breastfeeding. Sample size: considering 75% as the expected rate at the time of the infant hospital discharge and an absolute difference of 30% between groups, 95% confidence level (5% alpha error) and 80% power (20% beta error), 94 subjects would need to be enrolled (47 in each study arm). Expecting a 7.5% loss after randomization, 101 was the total number of subjects considered necessary to conduct the study; Test type: Superiority or Other; p = 0.06, Chi-squared; Risk Ratio (RR) = 1.22, 95% CI [0.99 to 1.51]

2. Secondary Outcome: Maternal Breastfeeding at 30 Days After Discharge
Description: as for outcome 1
Time Frame: At 30 days after the infant hospital discharge
Population: Analysis by intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 46 | 48
participants | 30 | 38
Statistical Analysis 1: Comparison: Control vs Music Therapy; Test type: Superiority or Other; p = 0.13, Chi-squared; Risk Ratio (RR) = 1.21, 95% CI [0.73 to 5.66]

3. Primary Outcome: Maternal Breastfeeding 7-15 Days After Discharge
Description: Maternal breastfeeding means: exclusive maternal breastfeeding, predominant maternal breastfeeding (maternal milk associated to other liquid, except formula) and continuous maternal breastfeeding (maternal milk associate to other food, including formula).
Time Frame: At the first follow-up visit (7-15 days after discharge)
Population: Analysis was by intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 46 | 48
participants | 32 | 42
Statistical Analysis 1: Comparison: Control vs Music Therapy; Null hypothesis: Music therapy does not increase the rate of maternal breastfeeding. Sample size: considering 75% as the expected rate at the time of the first follow-up visit and an absolute difference of 30% between groups, 95% confidence level (5% alpha error) and 80% power (20% beta error), 94 subjects would need to be enrolled (47 in each study arm). Expecting a 7.5% loss after randomization, 101 was the total number of subjects considered necessary to conduct the study; Test type: Superiority or Other; p = 0.03, Chi-squared; Risk Ratio (RR) = 1.26, 95% CI [1.01 to 1.57]

4. Secondary Outcome: Maternal Breastfeeding at 60 Days After Discharge
Description: as for outcome 1
Time Frame: At 60 days after the infant hospital discharge
Measure: Number; unit: participants
Arm/Group | Control | Music Therapy
Number analyzed (Participants) | 46 | 48
participants | 27 | 36
Statistical Analysis 1: Comparison: Control vs Music Therapy; Test type: Superiority or Other; p = 0.09, Chi-squared; Risk Ratio (RR) = 1.28, 95% CI [0.95 to 1.71]

ADVERSE EVENTS:
Arm/Group | Control | Music Therapy
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes